CLINICAL TRIAL: NCT02466477
Title: A Three-arm, Parallel Group, Multicentre, Double-blind, Randomized Controlled Trial Evaluating the Impact of GeneSight Psychotropic and Enhanced-GeneSight Psychotropic, on Response to Psychotropic Treatment in Outpatients Suffering From a Major Depressive Disorder (MDD) and Having Had - Within the Current Episode - an Inadequate Response to at Least One Psychotropic Medication Included in GeneSight Psychotropic
Brief Title: Pharmacogenomic Decision Support With GeneSight Psychotropic to Guide the Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assurex Health Inc. (Industry)
Collaborators: Programs for Assessment of Technology in Health Research Institute (Other); Centre for Addiction and Mental Health (Other); Genome Canada (Other); Assurex Health Ltd. (Unknown); Mars Excellence in Clinical Innovation and Technology Evaluation (Other)
Responsible Party: Principal Investigator, Ana Gugila, Sponsor, Assurex Health Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXCITE-013304-ARX1009.PTL
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Depressive Disorder, Major; Depression; Depressive Disorder
Keywords: Pharmacogenomic; Pharmacogenomic Testing; Pharmacogenomics; Genetic Testing; Genetics; Major Depressive Disorder; GeneSight; Enhanced GeneSight; Psychotropic
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GeneSight Psychotropic (GEN) (Experimental): The GeneSight Psychotropic (GEN) product is a pharmacogenomic decision support tool that helps clinicians to make informed, evidence-based decisions about proper drug selection. More specifically, patients are tested for clinically important genetic variants of multiple pharmacokinetic and pharmacodynamic genes that affect a patient's ability to metabolize, tolerate or respond to medications.
  Interventions: Genetic: GeneSight Psychotropic (GEN)
- Enhanced-GeneSight Psychotropic (E-GEN) (Experimental): The current GEN test lacks predictive genes for antipsychotic-induced weight gain (AIWG), a major complication of antipsychotic drug use. Therefore, the Enhanced-GeneSight Psychotropic (E-GEN), which is an enhanced version of the GEN test, was developed by incorporating 6 new genes (represented by 7 SNPs) that are predictive for AIWG, to those used in the GEN algorithm. An increasing risk level associated with AIWG is estimated by an increasing number of risk genotypes that a given patient possesses among the 7 SNPs.
  Interventions: Genetic: Enhanced-GeneSight Psychotropic (E-GEN)
- Treatment as Usual (TAU) (Active Comparator): The comparator chosen for this study provides a "real world" comparison of standard of care for patients who receive no pharmacogenomics guidance.
  Patients randomized to the TAU arm will also have their DNA collected and a pharmacogenomic-based interpretive report will be generated using GEN testing. However, this report will not be shared with the treating clinicians until completion at 12 months of the study. Therefore, patients in this arm will receive clinical treatment as usual, without the use or knowledge of genotyping results by their treating clinicians.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Genetic: GeneSight Psychotropic (GEN) — Patient DNA will be collected for all subjects and measured for variations in drug target genes and in drug metabolizing genes.Recommendations for optimal choices and dose adjustments for the 33 most commonly prescribed antidepressant and antipsychotic medications will be provided to subjects randomized to the GEN arm. This pharmacogenomic-based interpretive report will be provided to treating clinicians of patients in the GEN arm of the study, allowing clinicians to use the report to support their treatment decisions.
  Arms: GeneSight Psychotropic (GEN)
Genetic: Enhanced-GeneSight Psychotropic (E-GEN) — The E-GEN test incorporates into the existing GEN product new markers that are predictive of side effect of antipsychotic-induced weight gain (AIWG). The pharmacogenomic-based interpretive report from E-GEN will be provided to treating clinicians of patients in the E-GEN arm of the study, allowing clinicians to use the report to support their treatment decisions.
  Arms: Enhanced-GeneSight Psychotropic (E-GEN)
Other: Treatment as Usual (TAU) — Subjects randomized to the TAU arm will also require collection of patient DNA. A pharmacogenomic-based interpretive report will be generated from GEN, however, this report is not provided to the treating clinician until completion of the study.
  Arms: Treatment as Usual (TAU)

SUMMARY:
Evidence exists supporting the ability of genetic variations to influence patient drug response and side effects. Previous studies utilizing an open-label design have shown significant improvement in major depressive disorder (MDD) patient outcomes following use of the GeneSight Psychotropic (GEN) test. The first objective of this trial is to utilize a double-blinded, randomized clinical trial design to replicate previous findings of improvement in clinical outcomes in MDD subjects whose medication therapy was guided by GEN testing. Another objective is to determine the added benefit of Enhanced-GeneSight (E-GEN) compared to GEN for the pharmacogenomic guidance of treatment selections. Furthermore, this trial intends to develop an evidence-based case for the value of GEN and E-GEN to Canadian healthcare payers.

DETAILED DESCRIPTION:
The primary objectives of this study are 1) to compare the efficacy of GEN to treatment as usual (TAU) in improving response to psychotropic treatment in outpatients suffering from a MDD and having had - within the current episode - an inadequate response to at least one psychotropic medication included in GEN; and 2) to validate the utility of the new CAMH markers and demonstrate the superior predictive capabilities and greater clinical utility of E-GEN as compared to GEN.

This study is designed as a three-arm multi-centre, double-blind (participants and raters), randomized controlled trial to compare the clinical and economic outcomes of GEN, E-GEN and TAU for patients suffering from a MDD and having had - within the current episode - an inadequate response to at least one psychotropic medication included in GEN. Participants will be randomized in a 1:1:1 ratio to each of the three treatment arms. Recruitment will be 24 months. Follow-up will be 12 months.

Subjects will complete short diagnostic interviews specific to their clinical diagnosis, basic metabolic measures (eg. blood pressure, weight), and provide buccal swab samples for genetic analysis (the unanalyzed buccal swabs and associated DNA will be biobanked). During the first visit, blood and urine samples will be required for laboratory panel screening and blood biobanking. Subjects will be monitored over a one year period and clinical measures and healthcare resource utilization will be obtained. Treating clinicians in the GEN and E-GEN arms will receive an easy to implement report providing pharmacogenomic guidance for prescribing psychotropic medications to their patients.

The study will recruit subjects from 10 sites, stratified into 2 clusters. Nine study sites altogether will form one of the two stratified clusters. CAMH will constitute the tenth study site and the second stratified cluster.The sample size required for this study was calculated using effect size estimates drawn from a previous study conducted by Hall-Flavin et al [Pharmacogenetics Genomics 2013; 23(10)]. Assuming an effect size of 0.30 in HAM-D17 score favoring the treatment group, intra class coefficient between clusters of 20%, statistical power of 90%, an alpha level of 0.05, and an expected 16.7% rate of premature discontinuation by Week 8 (primary endpoint), a total of 570 subjects (i.e., 190 per treatment arm) are required to detect the same effect in this study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Suffer from a Major Depressive Episode meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria;
* Have had an inadequate response within the current episode to at least one psychotropic treatment in GEN. Inadequate response is defined as inadequate efficacy after 6 weeks of a psychotropic treatment or discontinuation of a psychotropic treatment due to adverse events (AEs) or intolerability;
* Have each a score on the 16-item Clinician Quick Inventory of Depressive Symptomatology (QIDS-C16) and 16-item Self-Report Quick Inventory of Depressive Symptomatology (QIDS-SR16) rating scales ≥ 11;
* Be able to understand the requirements of the study and provide written informed consent to participate in this study;
* Agree to abide by the study protocol and its restrictions and be able to complete all aspects of the study, including all visits and tests.

Exclusion Criteria:

* Patients posing a serious suicidal risk and/or in need of immediate hospitalization as judged by the Investigator;
* Patients with a diagnosis of Bipolar I or II disorder;
* Patients with a current Axis I diagnosis of:

  * Delirium
  * Dementia
  * Amnestic and/or other cognitive disorder
  * Schizophrenia or other psychotic disorder;
* Patients having experienced hallucinations, delusions, or any psychotic symptomatology within the current depressive episode or during prior depressive episodes;
* Patient is currently in an inpatient facility;
* Patients with a history of hypothyroidism unless taking a stable dose of thyroid medication and asymptomatic or euthyroid for at least 6 months;
* Patients who meet DSM-IV-TR criteria for any significant current substance use disorder;
* Patients with:

  * hepatic insufficiency (three times the upper limit of normal (ULN) for aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)); liver transplant recipient; cirrhosis of the liver;
  * malignancy (except basal cell carcinoma) and/or chemotherapy within 1 year prior to screening; malignancy more than 1 year prior to screening must have been local and without metastasis and/or recurrence, and if treated with chemotherapy, without nervous system complications;
  * significant unstable medical condition or life threatening disease with - need for therapies that may obscure the results of treatment and/or of the study;
* Participation in another clinical trial within 30 days of the screening visit;
* Anticipated inability to attend scheduled study visits;
* Patients who in the judgment of the Investigator may be unreliable or uncooperative with the evaluation procedure outlined in this protocol;
* Patients with a history of prior pharmacogenomic testing;
* Any change in psychotropic medication (including change in dosage) between screening and baseline;
* Patients currently receiving electroconvulsive therapy (ECT), deep brain stimulation (DBS) or transcranial magnetic stimulation (TMS) treatments, or currently scheduled to receive maintenance treatments of ECT, DBS, or TMS during the course of the study;
* Patients who self-report to be pregnant or lactating;
* Patients with a history of gastric bypass surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms as assessed by the 17-item Hamilton Depression (HAM-D17) score | From baseline to Week 8
  Mean change in the 17-item Hamilton Depression (HAM-D17) score from baseline to Week 8 of the study

SECONDARY OUTCOMES:
Change in depressive symptoms as assessed by the 16-Item Clinician Quick Inventory of Depressive Symptomatology (QIDS-SR16) | Baseline, Weeks 8 and 12, and Month 12
Change in depressive symptoms as assessed by the 9-Item Patient Health Questionnaire (PHQ-9) | Baseline, Weeks 8 and 12, and Month 12
Change in anxiety symptoms as assessed by theGeneralized Anxiety Disorder 7-Item (GAD-7) Scale | Baseline, Weeks 8 and 12, and Month 12
Change in severity of illness as assessed by the Clinical Global Impression of Severity (CGI-S) | Baseline, Week 12 and Month 12
Change in global improvement as assessed by the Clinical Global Impression of Improvement (CGI-I) | Week 12, and Month 12
Change in global therapeutic benefit and global severity of side effects as assessed by the Clinical Global Impression Efficacy Index | Week 12 and Month 12
Changes to initial prescribing based on availability of pharmacogenomic data | Screening and Baseline
Response rates to psychotropic medication | Baseline, Weeks 8 and 12, Months 6, 9 and 12
  A responder is defined as a participant with 50% decrease in HAM-D17 score from baseline.
Remission rates | Baseline, Weeks 8 and 12, Months 6, 9 and 12
  A remitter is defined as a participant with HAM-D17 score equal or less that 7.
Time to response | Baseline, Weeks 8 and 12, Months 6, 9 and 12
Time to remission | Baseline, Weeks 8 and 12, Months 6, 9 and 12
Change in psychotropic medication side effects as assessed by the Udvalg for Kliniske Undersogeler (UKU) Side Effect Rating Scale | Baseline, Weeks 8 and 12, and Month 12
Change in global measure of side effects (frequency, intensity, and burden domains) as assessed by the Frequency, Intensity, and Burden of Side Effects Ratings (FIBSER) | Baseline, Weeks 8 and 12, and Month 12
Weight gain | Baseline, Weeks 8 and 12, and Month 12
  Subject's weight
Waist-to-hip ratio | Baseline, Weeks 8 and 12, and Month 12
  Subject's waist and hip measurements
Change in health related quality of life as assessed by the EuroQol (EQ-5D-5L) | Baseline, Week 12, Months 6, 9 and 12
Change in health related quality of life as assessed by the Short Form (36) Health Survey (SF-36) | Baseline, Week 12, Months 6, 9 and 12
Pharmacogenetics in Psychiatry Follow-up Questionnaire (PIPFQ) | Baseline, when prescription changes are made (expected average of every 4 weeks), and Month 12
  The PIPFQ is a questionnaire developed by CAMH to evaluate each physician's attitude and experience to pharmacogenomic testing. Information is solicited from the physician on three different domains: the processing of the physician's last referral, the contact and outcome of the physician's patient, and the physician's perspective on the future of genetic studies in psychiatric drug treatment.
Healthcare resource utilization (Composite measure of healthcare costs): physician visits, hospital utilization, emergency department visits, medication use, and laboratory tests | Baseline, Weeks 8 and 12, Months 6, 9 and 12
Productivity losses (measured as economic costs) | Baseline, Weeks 8 and 12, Months 6, 9 and 12

CONTACTS AND LOCATIONS:
Overall Officials: James L Kennedy, MD, Principal Investigator — Centre for Addiction and Mental Health; Bryan Dechairo, PhD, Principal Investigator — Assurex Health Inc.
Locations (14):
- Canada (14):
  - Chatham-Kent Clinical Trials Research Center, Chatham, Ontario
  - Hamilton Community Health Centre Family Health Organization, Hamilton, Ontario
  - Hamilton Medical Research Group, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton (SJHH), Hamilton, Ontario
  - Milestone Research, London, Ontario
  - London Health Sciences Centre, London, Ontario
  - Parkwood Institute, London, London, Ontario
  - Hopital Montfort, Ottawa, Ontario
  - Thornhill Medical Centre, Thornhill, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Sinai Health System, Toronto, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
  - Manna Research, Toronto, Ontario

REFERENCES:
- [Derived] Tiwari AK, Zai CC, Altar CA, Tanner JA, Davies PE, Traxler P, Li J, Cogan ES, Kucera MT, Gugila A, Braganza N, Emmerson H, Zai G, Muller DJ, Levitan R, Kloiber S, Daskalakis ZJ, Frey BN, Bowen JM, Tarride JE, Tytus R, Chandrasena R, Voudouris N, Taylor VH, Tempier R, Sharma V, Vasudev A, Dzongowski P, Pliamm L, Greenspoon T, Dechairo BM, Kennedy JL. Clinical utility of combinatorial pharmacogenomic testing in depression: A Canadian patient- and rater-blinded, randomized, controlled trial. Transl Psychiatry. 2022 Mar 14;12(1):101. doi: 10.1038/s41398-022-01847-8. PMID 35288545

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT02466477/SAP_000.pdf
  • Study Protocol (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT02466477/Prot_001.pdf